CLINICAL TRIAL: NCT04272996
Title: Endovascular Embolization for Chronic Subdural Hematomas Following Surgical Evacuation
Acronym: endovascular
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Augusta University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1496700-3
Record Dates: First submitted 2020-02-11; First posted 2020-02-17 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Chronic SDH and the Efficacy of Embolization
Keywords: subdural hematoma; embolization; middle meningeal artery
MeSH Terms: conditions — Hematoma, Subdural | interventions — Craniotomy

STUDY DESIGN:
Intervention Model Description: The control group (surgery) would only receive surgical evacuation of a hematoma using current standard of care. The treatment group (surgery plus) would receive surgical evacuation followed by endovascular embolization of the middle meningeal vessels using current standard of care. We will directly compare these two treatment modalities to obtain class I evidence on the efficacy of embolization for treatment of chronic subdural hematomas.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- surgery alone (Other): craniotomy for SDH evacuation
  Interventions: Procedure: Craniotomy only
- Surgery plus embolization (Active Comparator): surgery for evacuation of SDH followed by embolization of middle meningeal vessel
  Interventions: Procedure: Craniotomy + Endovascular embolization of the middle meningeal vessels

INTERVENTIONS:
Procedure: Craniotomy only — evacuation of SDH
  Other Names: Craniotomy alone
  Arms: surgery alone
Procedure: Craniotomy + Endovascular embolization of the middle meningeal vessels — evacuation of SDH + Embolization of middle meningeal vessels using standard techniques.
  Arms: Surgery plus embolization

SUMMARY:
This study is designed to evaluate the effectiveness of endovascular embolization of middle meningeal artery following evacuation of subdural hematomas (SDHs) to assess rate of recurrence. The historical standard for treatment of subdural hematomas has been surgical evacuation through burr holes or craniotomies. Many of these patients are elderly patients who are high risk surgical candidates. A major concern is SDH recurrence.

Recurrences require frequent imaging, and will lead to increased length of hospital stay, increased morbidity,and re-operations. There are increasing number of reports that suggest that a less invasive approach such as endovascular embolization of the middle meningeal artery using standard endovascular materials and techniques may reduce the risk of recurrence. The reported outcomes in the current literature have been very positive when endovascular embolization has been used without surgery or as an adjuvant to surgery. However, there have been no studies directly comparing endovascular embolization following surgical evacuation to assess if this technique can actually reduce the complications of SDHs listed above. The investigators propose to study this treatment process by randomly assigning patients who have undergone surgical evacuation of SDHs into a control and treatment group. The control group will receive standard surgical evacuation of the hematoma. The study group will receive surgical evacuation followed by endovascular embolization.

DETAILED DESCRIPTION:
The historical standard for treatment of chronic subdural hematomas (SDH) has been through surgical evacuation through burr holes or craniotomies. Many of these patients are elderly patients who are high risk surgical candidates. Unfortunately given the pathophysiology of SDHs there is a high rate of recurrence ranging 5-30% in the literature necessitation frequent imaging, increased length of hospital stay, increased morbidity, and increased rate of reoperations. A more novel and less invasive approach has been used to treat SDHs in this patient population. There are increasing reports of endovascular embolization of the middle meningeal artery using a less invasive endovascular approach for SDHs. The reported outcomes in literature have been very positive when endovascular embolization has been used without surgery or as an adjuvant to surgery. These reports include case series and retrospective reviews. There have been no studies directly comparing endovascular embolization following surgical evacuation to assess if this technique can actually benefit patients with chronic SDHs. The investigators propose to study this treatment process by randomly assigning patients who have undergone surgical evacuation of SDHs through burr holes into a control and treatment group. The control group (surgery) would only receive surgical evacuation of the hematoma using current standard of care. The treatment group (surgery plus) would receive surgical evacuation followed by endovascular embolization of the middle meningeal vessels using current standard of care. We will directly compare these two treatment modalities to obtain class I evidence on the efficacy of embolization for treatment of chronic subdural hematomas.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18-90 with chronic SDH
* Patients that require surgical evacuation of SDH following assessment by a neurosurgeon
* Glasgow Coma Scale (GCS) >6
* Modified Rankin Scale (mRs) <5

Exclusion Criteria:

* Patients < 18 or >90 years of age
* Pregnancy
* Patients with extensive multisystem trauma requiring multidisciplinary surgical interventions
* Chronic renal insufficiency with creatinine >1.8
* GCS <6
* mRs >4
* Genetic bleeding disorder
* Liver failure
* Coagulopathy
* Patients unable to consent who do not have an LAR available

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
SDH recurrence | 3 months
  Radiographic assessment of SDH recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Fernando L. Vale, M.D., Principal Investigator — Medical College of Georgia-Augusta University
Locations (1):
- Augusta University, Augusta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sahyouni R, Goshtasbi K, Mahmoodi A, Tran DK, Chen JW. Chronic Subdural Hematoma: A Historical and Clinical Perspective. World Neurosurg. 2017 Dec;108:948-953. doi: 10.1016/j.wneu.2017.09.064. Epub 2017 Sep 19. PMID 28935548
- [Result] Link TW, Boddu S, Paine SM, Kamel H, Knopman J. Middle Meningeal Artery Embolization for Chronic Subdural Hematoma: A Series of 60 Cases. Neurosurgery. 2019 Dec 1;85(6):801-807. doi: 10.1093/neuros/nyy521. PMID 30418606
- [Result] Ban SP, Hwang G, Byoun HS, Kim T, Lee SU, Bang JS, Han JH, Kim CY, Kwon OK, Oh CW. Middle Meningeal Artery Embolization for Chronic Subdural Hematoma. Radiology. 2018 Mar;286(3):992-999. doi: 10.1148/radiol.2017170053. Epub 2017 Oct 10. PMID 29019449
- [Result] Fiorella D, Arthur AS. Middle meningeal artery embolization for the management of chronic subdural hematoma. J Neurointerv Surg. 2019 Sep;11(9):912-915. doi: 10.1136/neurintsurg-2019-014730. Epub 2019 Feb 23. PMID 30798265

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-27): https://cdn.clinicaltrials.gov/large-docs/96/NCT04272996/Prot_SAP_000.pdf